CLINICAL TRIAL: NCT02089295
Title: An Open-label, Randomized, Single-dose, Three-way Crossover Study to Evaluate the Dose Proportionality of 5 Mg, 20 Mg and 40 Mg of PF-00345439 Formulation K Under Intermediate-fat Fed Conditions in Healthy Volunteers
Brief Title: Dose Proportionality Study Of PF-00345439 Formulation Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501035
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: dose proportionality; oxycodone
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single dose of 5 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment B (Experimental): Single dose of 20 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone
- Treatment C (Experimental): Single dose of 40 mg PF-00345439 under naltrexone block (50 mg of naltrexone administered by mouth 12 hours before, 30 minutes before, and 12 hours after study drug administration).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — One capsule of 5 mg PF-00345439 Formulation K, single dose, under fed conditions
  Arms: Treatment A
Drug: Oxycodone — One capsule of 20 mg PF-00345439 Formulation K, single dose, under fed conditions
  Arms: Treatment B
Drug: Oxycodone — One capsule of 40 mg PF-00345439 Formulation K, single dose, under fed conditions
  Arms: Treatment C

SUMMARY:
To evaluate the dose proportionality of 5 mg, 20 mg and 40 mg of PF 00345439 formulation under fed conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Concentration at time 24 hours (C24) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
Plasma Decay Half-Life (t1/2) | 0,0.5,1,2,3,4,5,6,8,10,12,16,24,36,48
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501035&StudyName=Dose%20Proportionality%20Study%20Of%20PF-00345439%20Formulation%20Under%20Fed%20Conditions